CLINICAL TRIAL: NCT01816815
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group Study in 60 Healthy Tubal-ligated Women Aged 18 to 45 Years Investigating the Pharmacodynamic Effects of 5 Different Doses (0.1 - 5 mg) BAY1002670 After Daily Oral Administration Over 84 Days
Brief Title: Study in Healthy Tubal Ligated Women to Evaluate Pharmacodynamics, Safety and Pharmacokinetics of BAY1002670
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 14723; 2011-001760-22 (EudraCT Number)
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Leiomyoma
Keywords: PK/PD; BAY1002670
MeSH Terms: conditions — Leiomyoma | interventions — vilaprisan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- BAY1002670 [0.1mg] (Experimental): 0.1 mg BAY1002670, oral administration, four tablets to be taken daily, 84 consecutive days
  Interventions: Drug: BAY1002670
- BAY1002670 [0.5mg] (Experimental): 0.5 mg BAY1002670, oral administration, four tablets to be taken daily, 84 consecutive days
  Interventions: Drug: BAY1002670
- BAY1002670 [1.0mg] (Experimental): 1.0 mg BAY1002670, oral administration, four tablets to be taken daily, 84 consecutive days
  Interventions: Drug: BAY1002670
- BAY1002670 [2.0mg] (Experimental): 2.0 mg BAY1002670, oral administration, four tablets to be taken daily, 84 consecutive days
  Interventions: Drug: BAY1002670
- BAY1002670 [5.0mg] (Experimental): 5.0 mg BAY1002670, oral administration, four tablets to be taken daily, 84 consecutive days
  Interventions: Drug: BAY1002670
- Placebo (Placebo Comparator): Placebo for BAY1002670, oral administration, four tablets to be taken daily, 84 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1002670
  Arms: BAY1002670 [0.1mg]; BAY1002670 [0.5mg]; BAY1002670 [1.0mg]; BAY1002670 [2.0mg]; BAY1002670 [5.0mg]
Drug: Placebo
  Arms: Placebo

SUMMARY:
Effects of BAY1002670 on bleeding pattern: non-bleeding rate; on endometrium; on ovarian function; return of menstrual bleeding after treatment; safety and tolerability; PK/PD (pharmacokinetic/pharmacodynamic) relationship

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects
* Sterilized by tubal ligation
* Age 18-45 years
* Body mass index (BMI) at screening: ≥ 18 and ≤ 32 kg/m²
* At least 3 consecutive regular menstrual cycles with a cycle length of 24 - 35 days before first screening examination according to the subject's history
* Absence of clinically relevant abnormal findings in the pre-treatment endometrial biopsy

Exclusion Criteria:

* Regular use of medicines (incl. anabolics)
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Amenorrhea for more than 3 months within the last 6 months before the first screening examination
* Lacking suitability for frequent transvaginal ultrasonography (TVU) examinations
* Clinically relevant findings (e.g. blood pressure, electrocardiogram [ECG], physical and gynecological examination, laboratory examination)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Non-bleeding rate (i.e. women without bleeding from treatment day 9 until the end of treatment) | After three months

SECONDARY OUTCOMES:
Return of menstrual bleeding after treatment | Up to two months after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- Antwerp, Belgium
- Germany (3):
  - Neu-Ulm, Bavaria
  - Neuss, North Rhine-Westphalia
  - Berlin, State of Berlin
- Belfast, Belfast, United Kingdom

REFERENCES:
- [Derived] Schutt B, Kaiser A, Schultze-Mosgau MH, Seitz C, Bell D, Koch M, Rohde B. Pharmacodynamics and safety of the novel selective progesterone receptor modulator vilaprisan: a double-blind, randomized, placebo-controlled phase 1 trial in healthy women. Hum Reprod. 2016 Aug;31(8):1703-12. doi: 10.1093/humrep/dew140. Epub 2016 Jun 10. PMID 27288475